CLINICAL TRIAL: NCT06281561
Title: Effect of Intranasal Dexmedetomidine Premedication on Sleep Disturbance After General Anaesthesia
Brief Title: Dexmedetomidine Premedication for Post-anaesthesia Sleep Disturbance
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Yang Bin, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FirstAHXiamenU-YB
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Sleep Disturbance
Keywords: Sleep Disturbance; Dexmedetomidine; Anesthesia; propofol
MeSH Terms: conditions — Parasomnias | interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Nasal spray with nomal saline before anesthesia
  Interventions: Drug: Normal Saline
- Dexmedetomidine (Experimental): Nasal spray with dexmedetomidine before anesthesia
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Normal Saline — Female patients undergoing hysteroscopy receive nasal spray with normal saline before anesthesia
  Arms: Control
Drug: Dexmedetomidine — Female patients undergoing hysteroscopy receive nasal spray with dexmedetomidine before anesthesia
  Arms: Dexmedetomidine

SUMMARY:
The goal of this clinical trial is to learn about the effect of preoperative nasal spry with dexmedetomidine on postoperative sleep disturbance in young to middle-aged women undergoing hysteroscopy. The main questions it aims to answer are:1) what is the incidence of postoperative sleep disturbance in unisex patients who receive propofol anesthesia. 2) The preventive effect of preanesthesia nasal spray dexmedetomidine on postoperative sleep disturbance.

Participants will receive total intravenous propofol anaesthesia after dexmedetomidine nasal spray. Sleep quality will be monitored by using a Wearable devices and the PSQI which was used to assess sleep quality 1,2 days before the surgery and 1,3,7 days after surgery.

Researchers will compare the effects of 0.2 or 0.5 ug/kg dexmedetomidine to see if it help improve postanesthesia sleep quality.

DETAILED DESCRIPTION:
General anesthesia induces a drug-dependent state of unconsciousness and disrupts the normal 90-minute cycles of non-REM and REM sleep, resulting in significant suppression of physiological sleep during the postoperative period. This can lead to complications such as daytime fatigue, anxiety, pain, and a significant impact on mental and cognitive function. Currently, no effective interventions have been identified to prevent postoperative sleep disturbance. Dexmedetomidine induces a distinct sedative response, with a easy transition from sleep to wakefulness and deep sedation similar to natural sleep, while maintaining forebrain connectivity. This has clinical implications for reducing postoperative sleep disturbances by exploring optimal combinations of anaesthetic drugs.

In this study, all subjects meeting the inclusion criteria will be randomly assigned to one of three groups: Dexmedetomidine 0.2 ug/kg, Dexmedetomidine 0.5 ug/kg and normal saline as control group. All dexmedetomidine solutions were diluted to 0.6ml at different doses and prepared by a senior nurse who was not involved in the follow-up. All patients received no preoperative medication. On arrival in the waiting room, all patients were examined and received an intranasal spray of a total volume of 0.6ml 25 minutes before anesthesia. Patients, anesthetists, gynecologists and nurses were all blinded to group allocation. Patients received an intravenous cannula with lactated Ringer's solution. Heart rate, non-invasive blood pressure, electrocardiogram, and SpO2 and BIS were monitored during hysteroscopic procedures. Propofol was administered via the TCI infusion system using the Marsh pharmacokinetic parameters with a target plasma concentration of 3.2 ng/ml in three groups. The initial starting dose of propofol was based on the results of our pre-test and BIS. If the target was achieved and the BIS was <50, remifentanil was given at 1 ug/kg by pump and LMA was then placed. During the hysteroscopy, TCI was regulated according to the up and down method of Dixon, first described in 1965. TCI was upregulated by 0.1-0.2 when patients had a somatic response （unintended movement of the angelus orris or limbs） during cervical dilation. In the absence of limb movement, the subsequent target plasma concentration was reduced by 0.1 ng/ml. Emergency equipment and drugs were available at all times.

Early recovery will be evaluated in PACU and Later recovery will be measured using QoR-40 questionnaire. Sleep quality was monitored using a wearable device and assessed using the Pittsburgh Sleep Quality Index questionnaire 1-2 days before surgery and 1, 3, and 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1.Patients undergoing hysteroscopy in the hospital;2. American Society of Anesthesiologists Classification (ASA) I-II;3.No significant cardiovascular disease, liver, and kidney function within normal limits;4.Fully informed about the study and willing to participate by signing the informed consent form.

Exclusion Criteria:

1. ASA III-IV, severe cardiovascular disease, or poor physical condition;2. History of mental illness;3. History of sedative or antipsychotic drug use (neuroinhibitors, anxiolytics, antidepressants, benzodiazepines) for any reason;4. History of sleep disorders or have night shifts;5. Surgical complications (bleeding, reoperation, meningitis);6. Nasal deformity or nasal trauma.

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sleep quality at after intervention | 1-2 day before and 7 days after anesthesia exposure
  Wearable devices continuously records Night sleep duration, deep sleep proportion, light sleep proportion, rapid eye movement (REM) proportion, deep sleep continuity, waking times, and breathing quality.All these parameters are registered and combined in a report that indicates the degree of quality of the person's sleep as good, fair or poor.
Pittsburgh sleep quality index(PSQI) | 1 day or 2 days before anesthesia exposure and 1, 3, and 7 days after anesthesia exposure.
  Total scores range from 0 to 21, with higher scores indicating worse sleep quality. PSQI≥8 was defined as sleep disorder.

SECONDARY OUTCOMES:
Early recovery evaluated by Aldrete rating scale | Post anesthesia care unit time
  The total score is 10 points. Higher scores indicate better rehabilitation. When the patient's score was > 9, the patient could be considered for transfer out of PACU
Later Recovery evaluated by QoR-40 questionnaire | QoR-40 score on the third day after surgery
  The maximum total score is 200, with higher scores indicating better recovery quality

CONTACTS AND LOCATIONS:
Overall Officials: BIN YANG, Principal Investigator — The First Affiliated Hospital of Xiamen University

IPD SHARING:
Plan to Share IPD: Yes
We expect to release the original data on the ResMan original data sharing platform （IPD sharing platform）.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: February 2025

REFERENCES:
- [Background] Wang X, Hua D, Tang X, Li S, Sun R, Xie Z, Zhou Z, Zhao Y, Wang J, Li S, Luo A. The Role of Perioperative Sleep Disturbance in Postoperative Neurocognitive Disorders. Nat Sci Sleep. 2021 Aug 6;13:1395-1410. doi: 10.2147/NSS.S320745. eCollection 2021. PMID 34393534
- [Background] Purcell KF, Scarcella N, Chun D, Holland C, Stauffer TP, Bolognesi M, Lachiewicz P. Treating Sleep Disorders After Total Hip and Total Knee Arthroplasty. Orthop Clin North Am. 2023 Oct;54(4):397-405. doi: 10.1016/j.ocl.2023.05.008. Epub 2023 Jul 11. PMID 37718079
- [Result] Yu S, Xiong Y, Lu G, Xiong X. Effects of Preoperative Sleep Disorders on Anesthesia Recovery and Postoperative Pain in Patients Undergoing Laparoscopic Gynecological Surgery under General Anesthesia. Mediators Inflamm. 2022 Dec 15;2022:7998104. doi: 10.1155/2022/7998104. eCollection 2022. PMID 36570021
- [Result] Jia X, Song Y, Li Z, Yang N, Liu T, Han D, Sun Z, Shi C, Zhou Y, Shi J, Liu Y, Guo X. Melatonin regulates the circadian rhythm to ameliorate postoperative sleep disorder and neurobehavioral abnormalities in aged mice. CNS Neurosci Ther. 2024 Mar;30(3):e14436. doi: 10.1111/cns.14436. Epub 2023 Sep 22. PMID 37736695
- [Result] Shi Y, Sun Q, Wang Y, Chen C, Jin J, Wang W, Lu Y, Hua Y, Liu J, Bian J, Yi Z. Can dexamethasone improve postoperative sleep and postoperative delirium in elderly patients undergoing robot-assisted laparoscopic radical prostatectomy? Protocol for a prospective, randomized, double-blind, controlled study. Trials. 2023 Aug 8;24(1):505. doi: 10.1186/s13063-023-07521-8. PMID 37550718
- [Result] Zhang Y, Tan SL, Du J, Chen Y, Jia J, Feng JG, Liu KX, Zhou J. Dexmedetomidine alleviates neuroinflammation, restores sleep disorders and neurobehavioral abnormalities in rats with minimal hepatic encephalopathy. Int Immunopharmacol. 2021 Jul;96:107795. doi: 10.1016/j.intimp.2021.107795. Epub 2021 May 24. PMID 34162157
- [Result] De Zen L, Divisic A, Molinaro G, Solidoro S, Barbi E. Dexmedetomidine at Home for Intractable Dystonia and Insomnia in Children With Special Needs: A Case Series. J Pain Symptom Manage. 2023 Dec;66(6):e653-e657. doi: 10.1016/j.jpainsymman.2023.07.018. Epub 2023 Aug 5. PMID 37544550
- [Derived] Li X, Yan L, Wang L, Chen H, Yang B. Study on the preventive effect of dexmedetomidine on anesthetic associated sleep disturbance in young to middle-aged female patients undergoing hysteroscopy: a study protocol for a crossover randomized controlled trial. Trials. 2024 Jul 15;25(1):480. doi: 10.1186/s13063-024-08311-6. PMID 39010171